CLINICAL TRIAL: NCT00876044
Title: A Randomized, Double-Blind, Placebo-controlled Study Comparing Aflibercept Versus Placebo on the QTc Interval in Cancer Patients Treated With Docetaxel
Brief Title: A Study to Evaluate the Effects of Aflibercept on QTc Interval in Cancer Patients
Acronym: QUTIE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TES10897; EudraCT:2008-006796-80
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 4 mg/kg every 2 weeks
  Interventions: Drug: aflibercept (AVE0005)
- 2 (Placebo Comparator): matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aflibercept (AVE0005) — Intravenous route
  Arms: 1
Drug: placebo — Intravenous route
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the effects of aflibercept on the QTc interval in cancer patients.

Secondary objectives are to evaluate the effects of aflibercept on other electrocardiogram (ECG) parameters, clinical safety and pharmakokinetic (PK) parameters.

DETAILED DESCRIPTION:
All patients receive background treatment with docetaxel.

ELIGIBILITY:
Inclusion criteria:

* Solid malignancy, documented by pathologic report, for which treatment with single-agent docetaxel (administered every 3 weeks, at dose <75 mg/m2)is planned.
* Written informed consent

Exclusion criteria:

* Patient has received more than 2 prior lines of cytotoxic-containing chemotherapy
* Conditions with screening ECG repolarization difficult to interpret, or showing significant abnormalities. This includes, but is not limited to: high degree AV block, pace-maker, atrial fibrillation or flutter
* QTcF >480 msec on screening ECG

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
ECG parameters (QTcF interval) | Cycle 1 and Cycle 3

SECONDARY OUTCOMES:
Other ECG parameters | Cycle 1 and Cycle 3
Clinical safety (adverse events, serious adverse events) | maximum of 15 cycles
Pharmacokinetic parameters | Cycle 1 and Cycle 3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Maison-Blanche P, Vermorken JB, Goksel T, Machiels JP, Agarwala S, Rottey S, Daugaard G, Volovat C, Scheulen M, Sengelov L, Grecea D, Eniu A, Jager E, Meiri E, Cascinu S, Strumberg D, Demir G, Clemens M, Pinotti G, Nardi M, Guthrie T, Boelle E, Magherini E. A randomized, double-blind, placebo-controlled study to assess QTc interval prolongation of standard dose aflibercept in cancer patients treated with docetaxel. J Cardiovasc Pharmacol. 2013 Jun;61(6):495-504. doi: 10.1097/FJC.0b013e31828b73ff. PMID 23429593